CLINICAL TRIAL: NCT02808871
Title: Phase 2 Study of Safety, Tolerability and Efficacy of Pirfenidone in Patients With Rheumatoid Arthritis Interstitial Lung Disease (TRAIL1)
Brief Title: Phase ll Study of Pirfenidone in Patients With RAILD (TRAIL1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Hilary J. Goldberg, M.D., Attending Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017p000062
Record Dates: First submitted 2016-03-20; First posted 2016-06-22 (Estimated); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis Interstitial Lung Disease
Keywords: TRAIL1; TRAIL; Pirfenidone
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pirfenidone (Experimental): Pirfenidone 2403 mg/d for 52 weeks
  Interventions: Drug: Pirfenidone
- Placebo (Placebo Comparator): Placebo for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone three times daily (2403 mg) for 52 weeks
  Other Names: Esbriet
  Arms: Pirfenidone
Drug: Placebo — Placebo three times daily for 52 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to to assess the safety and tolerability of pirfenidone 2403 mg/day for the treatment of RA-associated interstitial lung disease.

DETAILED DESCRIPTION:
This is a phase 2, randomized, double blind, placebo controlled trial of pirfenidone for the treatment of RA associated interstitial lung disease. Approximately 270 subjects will be randomized to receive Pirfenidone 2403 mg per day or placebo in a 1:1 ratio. The primary outcome of this study is to assess the efficacy of pirfenidone 2403 mg/day versus placebo in patients with RA associated interstitial lung disease, as defined by progression free survival over the 52 weeks of treatment. Patients will receive blinded study treatment from the time of randomization until the Week 52 Visit.

Eligible patients aged 18 to 85 years must meet 2010 ACR/EULAR criteria for RA (Aletaha, Neogi et al. 2010) as well as RA-associated ILD, as determined by imaging and, when available, lung biopsy. Patients will be required to have a % predicted FVC ≥40 and % predicted DLCO or TLCO ≥30 at screening.

The dose of study treatment will be titrated over 14 days. Patients will receive a telephone assessment at Weeks 1 and 2, and visit the clinic at Weeks 4, 8, 13, 19, 26, 39, and 52. Subjects will have a follow up phone call 28 days after completion of the study drug. Patients should complete a compliance diary between visits. If patients discontinue study treatment for any reason before the end of the study, they should continue with all scheduled study procedures through Week 52. If subjects are unable to complete the study visits as scheduled, all efforts should be made to complete an early termination visit.

The primary outcome variable of this study will be progression free survival, defined as progression free from decline in FVC of 10% or greater during the 52 week study period.

More information can be found at www.ralung.org.

ELIGIBILITY:
Patients must fulfill all of the following criteria to be eligible for enrollment in the study:

1. Age 18 through 85 years, inclusive, at Screening
2. Probable or definite diagnosis of RA according to revised 2010 ACR/EULAR criteria, without evidence or suspicion of an alternative diagnosis that may contribute to their interstitial lung disease.
3. Diagnosis of ILD

   1. supported by clinically indicated HRCT, and when available, surgical lung biopsy (SLB), prior to Screening, and
   2. presence of fibrotic abnormality affecting more than 10% of the lung parenchyma, with or without traction bronchiectasis or honeycombing, on screening and confirmed by adjudicated HRCT prior to Baseline
4. No features supporting an alternative diagnosis on transbronchial biopsy, or SLB, if performed prior to Screening
5. Attainment of the following centralized spirometry criteria (based on local spirometry on standardized equipment and centralized quality controlled):

   1. percent predicted FVC ≥ 40% at Screening
   2. change in pre-bronchodilator FVC (measured in liters) between Visit 1 (Screening) and Visit 2 (Randomization) must be a <10% relative difference, calculated as: 100% * [absolute value (Visit 1 FVC - Visit 2 FVC) / Visit 1 FVC]
   3. percent predicted DLCO or TLCO ≥25 % at Screening
   4. Screening (Visit 1) pre-bronchodilator(BD) and Post-BD spirometry meets ATS quality criteria as determined by a central reviewer
   5. Baseline (Visit 2) Pre-BD spirometry meets ATS quality criteria as determined by the site Investigator or the central reviewer
6. Able to understand and sign a written informed consent form.
7. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, during the 52 week treatment period and for at least 118 days after the last dose of study drug.

   1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
   2. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
   3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
8. For men who are not surgically sterile: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

   1. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 118 days after the last dose of study drug.
   2. Men must refrain from donating sperm during this same period.

PARTICIPANT EXCLUSION CRITERIA

1. Not a suitable candidate for enrollment or unlikely to comply with the requirements of this study, in the opinion of the investigator
2. Cigarette smoking or vaping within 3 months of Screening or unwilling to avoid tobacco products throughout the study
3. History of clinically significant environmental exposure known to cause pulmonary fibrosis (PF), including but not limited to drugs (such as amiodarone), asbestos, beryllium, radiation, and domestic birds
4. Concurrent presence of the following conditions:

   1. Other interstitial lung disease, related to but not limited to radiation, drug toxicity, sarcoidosis, hypersensitivity pneumonitis, or bronchiolitis obliterans organizing pneumonia
   2. Medical history including Human Immunodeficiency Virus (HIV)
   3. Medical history of viral hepatitis (positive Hep A antibody in the absence of elevated liver enzymes is not an exclusion)
5. Concurrent presence of other pleuropulmonary manifestations of RA, including but not limited to rheumatoid nodular disease of the lung, pleuritis/pleural thickening, and obliterative bronchiolitis
6. Post-bronchodilator FEV1/FVC <0.65 at Screening
7. Presence of pleural effusion occupying more than 20% of the hemithorax on Screening HRCT
8. Clinical diagnosis of a second connective tissue disease or overlap syndrome (including but not limited to scleroderma, sjogren's, polymyositis/dermatomyositis, systemic lupus erythematosus but excluding Raynaud's phenomena)
9. Coexistent clinically significant COPD/emphysema or asthma in the opinion of the site principal investigator
10. Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis, urinary tract infection, or cellulitis. The infection should be resolved per PI assessment prior to enrollment. Any use of antibiotics must be completed 2weeks prior to the screening visit. Note that prophylactic antibiotics are not contraindicated or exclusionary
11. Any history of malignancy diagnosed within 5 years of screening, other than basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or low grade cervical carcinoma, and/or low grade prostate cancer.

    Criteria for low grade prostate cancer:
    * Patients with suspicion for prostate cancer based on PSA and/or DRE should have been evaluated by urology
    * Patients with NCCN very low risk prostate cancer (∙ T1c and Grade Group 1 (Gleason 6) and PSA <10 ng/mL and Fewer than 3 prostate biopsy fragments/cores positive, ≤50% cancer in each fragment/coreg and ∙ PSA density <0.15 ng/mL/g) can be monitored without intervention and enrolled in study.
    * Patients with NCCN low risk prostate cancer can be monitored on a case by case basis (T1-T2a and Grade Group 1 (Gleason 6) and ∙ PSA <10 ng/mL) and enrolled in study.
    * All other patients should be excluded.
12. History of LFT abnormalities as outlined below, or imaging, laboratory or other clinical information suggesting liver dysfunction, advanced liver disease or cirrhosis. Evidence of hepatic impairment that in the opinion of the investigator could interfere with drug metabolism or increase the risk of the known hepatotoxicity of study drug.

    Any of the following liver function abnormalities:
    1. Total bilirubin above the upper limit of normal (ULN), excluding patients with Gilbert's syndrome;
    2. Aspartate or alanine aminotransferase (AST/SGOT or AST/SGPT) > 3 X ULN;
    3. Alkaline phosphatase > 2.5 X ULN.
13. History of end-stage renal disease requiring dialysis
14. History of unstable or deteriorating cardiac disease, or unstable cardiac arrhythmia or arrhythmia requiring modification of drug therapy, myocardial infarction within the previous year, heart failure requiring hospitalization.
15. Any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of pirfenidone
16. History of alcohol or substance abuse in the past 2 years, at the time of Screening
17. Family or personal history of long QT syndrome
18. Any of the following test criteria above specified limits:

    1. Estimated glomerular filtration rate <30 mL/min/1.73m2
    2. ECG with a QTc interval >500 msec at Screening
19. Prior use of pirfenidone or known hypersensitivity to any of the components of study treatment
20. Use of any of the following therapies within 28 days before Screening and during participation in the study:

    1. Investigational therapy, defined as any drug that has not been approved for marketing for any indication in the country of the participating site
    2. Potent inhibitors of CYP1A2(e.g. fluvoxamine, enoxacin)
    3. Potent inducers of CYP1A2.
    4. Sildenafil (daily use). Note: intermittent use for erectile dysfunction is allowed
21. Introduction and/or modification of dose of corticosteroids or any cytotoxic, immunosuppressive, or cytokine modulating or receptor antagonist agent for the management of pulmonary manifestations of RA, within 3 months of screening, is an exclusion criterion for enrollment, with the exception of dose modification of systemic corticosteroids that are maintained at or below 20 mg prednisone daily or the equivalent.

    However, introduction and/or modification of dose of corticosteroids or any cytotoxic, immunosuppressive, or cytokine modulating or receptor antagonist agent for the management of extrapulmonary manifestations of RA is not an exclusion criterion for enrollment.
22. Any use of an approved anti-fibrotic medication within 28 days of screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan O. Rosas, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (33):
- United States (13):
  - University of Alabama Site at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Miami, Miami, Florida
  - Tulane Medical Center, New Orleans, Louisiana
  - John Hopkins Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah Health Care, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Australia (4):
  - Royal Brompton, Brisbane, Queensland
  - Royal Prince Alfred Hospital, Camperdown, Sydney
  - Melbourne Alfred Hospital, Melbourne, Victoria
  - The Prince Charles Hospital, Camperdown
- Canada (4):
  - University of Calgary Cummings School of Medicine, Calgary, Alberta
  - St. Paul's Hospital - Providence Health Care, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
- United Kingdom (12):
  - North Bristol NHS Trust Headquarters, Southmead Hospital, Bristol
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Royal Devon and Exeter NHS Foundation, Exeter
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Aintree University Hospitals NHS Foundation Trust, Liverpool
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust (South) Wythenshawe Hospita, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solomon JJ, Danoff SK, Woodhead FA, Hurwitz S, Maurer R, Glaspole I, Dellaripa PF, Gooptu B, Vassallo R, Cox PG, Flaherty KR, Adamali HI, Gibbons MA, Troy L, Forrest IA, Lasky JA, Spencer LG, Golden J, Scholand MB, Chaudhuri N, Perrella MA, Lynch DA, Chambers DC, Kolb M, Spino C, Raghu G, Goldberg HJ, Rosas IO; TRAIL1 Network Investigators. Safety, tolerability, and efficacy of pirfenidone in patients with rheumatoid arthritis-associated interstitial lung disease: a randomised, double-blind, placebo-controlled, phase 2 study. Lancet Respir Med. 2023 Jan;11(1):87-96. doi: 10.1016/S2213-2600(22)00260-0. Epub 2022 Sep 5. PMID 36075242
- [Derived] Solomon JJ, Danoff SK, Goldberg HJ, Woodhead F, Kolb M, Chambers DC, DiFranco D, Spino C, Haynes-Harp S, Hurwitz S, Peters EB, Dellaripa PF, Rosas IO; Trail Network. The Design and Rationale of the Trail1 Trial: A Randomized Double-Blind Phase 2 Clinical Trial of Pirfenidone in Rheumatoid Arthritis-Associated Interstitial Lung Disease. Adv Ther. 2019 Nov;36(11):3279-3287. doi: 10.1007/s12325-019-01086-2. Epub 2019 Sep 12. PMID 31515704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pirfenidone | Placebo
Started | 63 | 60
Completed | 52 | 51
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone | Placebo | Total
Number analyzed (Participants) | 63 | 60 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 18 | 45
  >=65 years | 36 | 42 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (8.2) | 68.1 (9.1) | 67.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 38 | 39 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 56 | 56 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 5 | 11
  United States | 25 | 23 | 48
  United Kingdom | 27 | 27 | 54
  Australia | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Any Element of the Composite Endpoint
Description: Number of participants who developed any element of the composite endpoint of decline in percent predicted FVC of 10% or greater or death.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 7 | 9

2. Secondary Outcome: Number of Participants With FVC Decline From Baseline of 10% or Greater
Description: Number of participants with decline from baseline in percent predicted FVC of 10% or greater during the study period.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 5 | 7

3. Secondary Outcome: Number of Participants With Progressive Disease
Description: Number of participants with progressive disease as defined by OMERACT: FVC% relative decline of >=10% or FVC% change in >=5< 10% and >=15% diffusing capacity (DLCO)
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 16 | 19

4. Secondary Outcome: Change in Absolute Value FVC Over the 52 Week Study Period
Description: Change from baseline to end of study in absolute value of FVC over the 52 week study period
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
ml | -66 (20) | -146 (20)

5. Secondary Outcome: Change in % Predicted FVC From Baseline to End of Study Over the 52 Week Study Period
Description: Change from baseline to end of study of percent predicted FVC over the 52 week study period
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
% predicted | -1.02 (0.51) | -3.21 (0.52)

6. Secondary Outcome: Time to Composite of Decline in FVC or Death
Description: Time to decline of 10% or greater in percent predicted FVC or death while on study
Time Frame: 52 weeks
Measure: Mean (Standard Error); unit: days
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
days | 349.5 (7.2) | 339.9 (10.2)

7. Secondary Outcome: Change in PRO of Dyspnea
Description: Change from Baseline to end of study in dyspnea, as measured by the Dyspnea 12 questionnaire - Total scores range from 0 to 36, with higher scores corresponding to greater severity.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
score | 0.45 (0.71) | 1.37 (0.72)

8. Secondary Outcome: All-cause Mortality
Description: Number of participants experiencing mortality due to all causes
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 2 | 3

9. Secondary Outcome: All Cause Hospitalization
Description: Number of participants requiring hospitalization for any cause
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Pirfenidone: Received pirfenidone
- Placebo: Received placebo
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 7 | 7

10. Secondary Outcome: Hospitalization for Respiratory Cause
Description: Number of participants requiring hospitalization for respiratory cause
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 2 | 5

11. Secondary Outcome: Acute Exacerbations Requiring Hospitalization
Description: Number of participants experiencing acute exacerbation requiring hospitalization
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 63 | 60
Participants | 1 | 2

12. Secondary Outcome: Treatment-emergent Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (AEs)
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 62 | 56

13. Secondary Outcome: Treatment-emergent Serious Adverse Events (SAEs)
Description: Number of participants with treatment-emergent serious adverse events (SAEs) in the as treated population
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 9 | 8

14. Secondary Outcome: Treatment-emergent/Treatment-related AEs
Description: Number of participants with treatment-emergent/treatment-related AEs
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 27 | 18

15. Secondary Outcome: Treatment-emergent/Treatment-related SAEs
Description: Number of participants with treatment-emergent/treatment-related SAEs
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 1 | 0

16. Secondary Outcome: AEs Leading to Early Discontinuation of Study Treatment
Description: Number of participants with AEs leading to early discontinuation of study treatment
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 15 | 6

17. Secondary Outcome: Treatment-emergent Death or Transplant
Description: Number of participants who experienced treatment-emergent death or transplant
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 2 | 4

18. Secondary Outcome: Treatment-emergent RA-ILD-related Mortality
Description: Number of participants who experienced treatment-emergent RA-ILD-related mortality
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 62 | 60
Participants | 1 | 0

19. Other Pre Specified Outcome: Disease Activity Score (DAS)
Description: Change from Baseline to end of study in Disease Activity Score (DAS)
Time Frame: 52 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: RAPID3 Score
Description: Change from baseline to end of study in Routine Assessment of Patient Index Data 3 (RAPID3) score
Time Frame: 52 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: Change from Baseline to end of study in Erythrocyte Sedimentation Rate (ESR)
Time Frame: 52 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: CRP
Description: Change from Baseline to end of study in C-Reactive Protein (CRP) 5. Candidate
Time Frame: 52 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Biomarker Expression
Description: Candidate biomarker expression in the peripheral blood of patients with RA-ILD over the 52 weeks of treatment
Time Frame: 52 weeks
Reporting Status: Not Posted

24. Other Pre Specified Outcome: HRCT Parameters
Description: Changes from Baseline to end of study in high resolution computed tomography (HRCT) parameters evaluated by quantitative functional imaging
Time Frame: 52 weeks
Reporting Status: Not Posted

25. Other Pre Specified Outcome: SGRQ
Description: Changes from Baseline to Week 13, 26, 39 and final visit in the St. George's Respiratory Questionnaire (SGRQ)
Time Frame: 52 weeks
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Dyspnea 12
Description: Changes from Baseline to Week 13, 26, 39 and final visit in Dyspnea 12 questionnaire
Time Frame: 52 weeks
Reporting Status: Not Posted

27. Other Pre Specified Outcome: LCQ
Description: Changes from Baseline to Week 13, 26, 39 and final visit in Leicester Cough Questionnaire (LCQ)
Time Frame: 52 weeks
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Patient Global Assessment
Description: Changes from Baseline to Week 13, 26, 39 and final visit in the Patient global assessment
Time Frame: 52 weeks
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Health Assessment Questionnaire
Description: Changes from Baseline to Week 13, 26, 39 and final visit in the Health assessment questionnaire
Time Frame: 52 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each participant was assessed for development of AE's from time of first dose of study drug through last study visit (56 weeks) or until withdrawal from study. Mean time period of AE monitoring per study subject was 51.5 weeks (SD 12.86).
Description: Adverse Events were monitored/assessed according to system/class without regard to the specific Adverse Event Term. Adverse events were measured in the as treated population.
Arm/Group | Pirfenidone | Placebo
All-Cause Mortality (participants affected / at risk) | 2/63 | 3/60
Serious Adverse Events (participants affected / at risk) | 10/62 | 11/60
Other Adverse Events (participants affected / at risk) | 62/62 | 56/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=62) | Placebo (N=60)
Cardiac (Cardiac disorders) | 3 | 0
Gastrointestinal (Gastrointestinal disorders) | 1 | 1
Immune System (Immune system disorders) | 1 | 0
Infections and Infestations (Infections and infestations) | 3 | 3
Musculoskeletal and Connective Tissue (Musculoskeletal and connective tissue disorders) | 0 | 2
Nervous System (Nervous system disorders) | 0 | 2
Respiratory, Thoracic and Mediastinal (Respiratory, thoracic and mediastinal disorders) | 2 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pirfenidone (N=62) | Placebo (N=60)
Blood and Lymphatic System (Blood and lymphatic system disorders) | 7 | 6
Cardiac (Cardiac disorders) | 12 | 9
Ear and Labyrinth (Ear and labyrinth disorders) | 5 | 2
Endocrine (Endocrine disorders) | 1 | 1
Eye (Eye disorders) | 8 | 4
Gastrointestinal (Gastrointestinal disorders) | 50 | 36
General (General disorders) | 37 | 28
Hepatobiliary (Hepatobiliary disorders) | 5 | 2
Immune System (Immune system disorders) | 4 | 3
Infections and Infestations (Infections and infestations) | 23 | 22
Injury, Poisoning and Procedural (Injury, poisoning and procedural complications) | 1 | 4
Investigations (Investigations) | 0 | 1
Metabolism and Nutrition (Metabolism and nutrition disorders) | 6 | 4
Musculoskeletal and Connective Tissue (Musculoskeletal and connective tissue disorders) | 30 | 23
Nervous System (Nervous system disorders) | 6 | 7
Psychiatric (Psychiatric disorders) | 5 | 2
Renal and Urinary (Renal and urinary disorders) | 2 | 5
Reproductive System and Breast (Reproductive system and breast disorders) | 1 | 1
Respiratory, Thoracic and Mediastinal (Respiratory, thoracic and mediastinal disorders) | 34 | 32
Skin and Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 20 | 15
Surgical and Medical Procedures (Surgical and medical procedures) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT02808871/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02808871/SAP_001.pdf